CLINICAL TRIAL: NCT05416632
Title: Diagnostic Accuracy of Hand Held Arthrometry and Clinical Tests for Diagnosing ACL Tears
Brief Title: Arthrometry and Clinical Tests for Diagnosing ACL Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SP0925
Record Dates: First submitted 2022-05-25; First posted 2022-06-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2023-03

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Tear
Keywords: Arthrometry; Lachmeter; Rolimeter
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Masking Description: Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arthrometer (Experimental)
  Interventions: Diagnostic Test: Athrometer

INTERVENTIONS:
Diagnostic Test: Athrometer — Arthrometer

SUMMARY:
Anterior cruciate ligament (ACL) tears are diagnosed by combining the patient's history and physical examination but clinical tests (e.g., Lachman, anterior drawer, and pivot shift) are less accurate within the first three weeks of injury. The Lever sign is a clinical test that has shown to have comparable diagnostic accuracy regardless of the time since injury, but this test has not been subjected to a randomised clinical trial and diagnostic values may be overestimated.

Imaging modalities (e.g., MRI) are utilised when clinical diagnosis is not clear but are expensive and delay diagnosis. Hand-held arthrometry is an instrument that can be used in the clinical setting to provide an immediate, objective measure of ACL laxity, but this device has not been adequately validated.

The first aim of this study is to determine the accuracy of hand-held arthrometry for diagnosing ACL tears following acute injury. A reliable and valid device could reduce healthcare costs and expedite appropriate treatment, thereby improving the management of patients following knee injury. The second aim of this study is to determine the diagnostic accuracy of the Lever sign test using a more robust study design than previously employed in other studies.

DETAILED DESCRIPTION:
Approximately 40-50% of patients that present with immediate knee swelling (within 2 hours) following injury have an anterior cruciate ligament (ACL) tear. Potential consequences of an ACL tear include further knee injury, post-traumatic osteoarthritis, and reduced quality of life, therefore prompt, accurate diagnosis is important to expedite treatment and mitigate these risks. Within the first three weeks of injury, clinical tests have lower diagnostic accuracy due to pain, swelling and patient guarding making it difficult to assess the integrity of the ACL with confidence.

Magnetic resonance imaging (MRI) is often performed following knee trauma, as immediate swelling is associated with significant knee injury. However, MRI is costly and can result in a significant delay in diagnosis due to the time it takes for the scan to be performed, reported and acted on. Hand-held arthrometers are clinical instruments that provide immediate, objective measurement of knee laxity, which can then be used to inform decision making. Previous research indicates a side-to-side difference in laxity >3mm is diagnostic for an ACL rupture, with <3mm indicating a partial tear, but this device has not been adequately evaluated in acute presentations. In addition, the accuracy of ACL tests has not been adequately evaluated using robust methodology (randomised control trial) so diagnostic values may have been previously overestimated.

The objective of this study is to determine the diagnostic accuracy of hand-held arthrometry in acute presentations (<3 weeks) using MRI as the reference standard and a prospective design. In addition, a blinded, randomised control trial will be conducted using known ACL- injured and non-injured patients (based on MRI results), to provide robust diagnostic accuracy values for clinical ACL tests.

The hypothesis is that hand-held arthrometry will have superior diagnostic accuracy to the Lachman values reported in the systematic review and meta-analysis of Sokal et al (Sn: 0.89, Sp: 0.62, LR+ 1.79, LR- 0.33). A second hypothesis is that the Lever sign diagnostic accuracy values will be inferior to those reported in the the SR and MA of Sokal et al (Sn: 0.83, Sp: 0.91, LR+ 9.66, LR- 0.18). If arthrometry provides a reliable and valid measure of knee laxity, the device could save significant costs and delays to diagnosis associated with MRI.

ELIGIBILITY:
Inclusion Criteria:

* History of knee injury (<3 weeks since trauma for the validity study) with immediate swelling (<2 hours) but no fracture on X-ray.
* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* No contraindications to arthrometer testing or MRI (see exclusion criteria).
* Healthy contralateral knee; no current or previous history of significant knee injury, or a history of previous minor injury that is symptomatic at the time of recruitment. No previous knee surgery.

Exclusion Criteria:

The participant may not enter the study if they are unable to provide written consent to study participation, or there are contraindications to arthrometer testing or MRI, including the following:

* History of chronic disease or disorder that may put the participants at risk because of participation in the study including non-united fractures, severe peripheral vascular disease, aneurysms, recent (<3 months) radiotherapy or chemotherapy, neurological disorders (e.g., Parkinson's disease), skin conditions at point of testing, severe osteoporosis, malignancy, rheumatoid arthritis.
* Patients with implanted surgical clips or other ferromagnetic material including shrapnel, metallic implants (excluding joint replacements >6 weeks since surgery), non-MRI compatible prosthetic heart valves, surgery within 6 weeks, pregnancy, patients with compromised thermoregulatory systems.
* History of chronic musculoskeletal disease or disorder in either leg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Accuracy reliability and validity of hand-held arthrometry. | 104 weeks
  Side to side differences in anterior tibial translation (measured in millimetres) using the arthrometer.

SECONDARY OUTCOMES:
To determine diagnostic accuracy of Lever sign test. | 104 weeks
  Dichotomous 'positive' or 'negative' ACL clinical test result.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Norris, Principal Investigator — Liverpool University Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Liverpool University Hospitals Nhs Foundation Trust, Liverpool, Merseyside
  - Aintree University Hospital NHS Foundation Trust, Liverpool, Merseyside

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbasi D, May MM, Wall EJ, Chan G, Parikh SN. MRI findings in adolescent patients with acute traumatic knee hemarthrosis. J Pediatr Orthop. 2012 Dec;32(8):760-4. doi: 10.1097/BPO.0b013e3182648d45. PMID 23147616
- [Background] Olsson O, Isacsson A, Englund M, Frobell RB. Epidemiology of intra- and peri-articular structural injuries in traumatic knee joint hemarthrosis - data from 1145 consecutive knees with subacute MRI. Osteoarthritis Cartilage. 2016 Nov;24(11):1890-1897. doi: 10.1016/j.joca.2016.06.006. Epub 2016 Jun 29. PMID 27374877
- [Background] Sarimo J, Rantanen J, Heikkila J, Helttula I, Hiltunen A, Orava S. Acute traumatic hemarthrosis of the knee. Is routine arthroscopic examination necessary? A study of 320 consecutive patients. Scand J Surg. 2002;91(4):361-4. doi: 10.1177/145749690209100410. PMID 12558087
- [Background] Filbay SR, Grindem H. Evidence-based recommendations for the management of anterior cruciate ligament (ACL) rupture. Best Pract Res Clin Rheumatol. 2019 Feb;33(1):33-47. doi: 10.1016/j.berh.2019.01.018. Epub 2019 Feb 21. PMID 31431274
- [Background] van Eck CF, van den Bekerom MP, Fu FH, Poolman RW, Kerkhoffs GM. Methods to diagnose acute anterior cruciate ligament rupture: a meta-analysis of physical examinations with and without anaesthesia. Knee Surg Sports Traumatol Arthrosc. 2013 Aug;21(8):1895-903. doi: 10.1007/s00167-012-2250-9. Epub 2012 Oct 20. PMID 23085822
- [Background] Hatcher J, Hatcher A, Arbuthnot J, McNicholas M. An investigation to examine the inter-tester and intra-tester reliability of the Rolimeter knee tester, and its sensitivity in identifying knee joint laxity. J Orthop Res. 2005 Nov;23(6):1399-403. doi: 10.1016/j.orthres.2005.06.003.1100230623. Epub 2005 Aug 3. PMID 16084050
- [Background] Decary S, Ouellet P, Vendittoli PA, Roy JS, Desmeules F. Diagnostic validity of physical examination tests for common knee disorders: An overview of systematic reviews and meta-analysis. Phys Ther Sport. 2017 Jan;23:143-155. doi: 10.1016/j.ptsp.2016.08.002. Epub 2016 Aug 5. PMID 27693100
- [Background] Muellner T, Bugge W, Johansen S, Holtan C, Engebretsen L. Inter- and intratester comparison of the Rolimeter knee tester: effect of tester's experience and the examination technique. Knee Surg Sports Traumatol Arthrosc. 2001 Sep;9(5):302-6. doi: 10.1007/s001670100225. PMID 11685363
- [Background] Sokal PA, Norris R, Maddox TW, Oldershaw RA. The diagnostic accuracy of clinical tests for anterior cruciate ligament tears are comparable but the Lachman test has been previously overestimated: a systematic review and meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2022 Oct;30(10):3287-3303. doi: 10.1007/s00167-022-06898-4. Epub 2022 Feb 12. PMID 35150292
- [Derived] Norris R, Price A, Byrne J, Pulford S, van Melick N, Maddox TW, Boswell W, Kerin C, Oldershaw RA. The Lever Sign Test Demonstrates Limited Clinical Utility for Diagnosing Full-Thickness Anterior Cruciate Ligament Tears After a Traumatic Knee Injury. Orthop J Sports Med. 2025 May 14;13(5):23259671251334775. doi: 10.1177/23259671251334775. eCollection 2025 May. PMID 40376390